CLINICAL TRIAL: NCT00790647
Title: Phase II Trial of High-dose Melphalan and Bortezomib and Stem Cell Transplantation in Patients With AL Amyloidosis
Brief Title: Melphalan, Bortezomib, and Stem Cell Transplant in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Vaishali Sanchorawala, Principal Investigator, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000618857; BUMC-H-27277 (Other: Boston University Medical Center IRB)
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Bortezomib; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplant with Bortezomib and Melphalan (Experimental): Mobilization with Filgrastim Stem Cell Collection Bortezomib Melphalan Stem Cell infusion
  Interventions: Biological: filgrastim; Drug: bortezomib; Drug: melphalan; Procedure: Stem Cell Infusion

INTERVENTIONS:
Biological: filgrastim — 16 mcg/kg daily beginning 3 days before stem cell collection through day before final stem cell collection
  Other Names: Growth-Colony Stimulating Factor, neupogen
Drug: bortezomib — 1.0 mg/m2/dose D -6, D-3, D +1, D + 4
  Other Names: velcade
Drug: melphalan — 100 mg/m2/dose D -2, D -1
  Other Names: alkeran
Procedure: Stem Cell Infusion — infusion of previously collected autologous stem cells

SUMMARY:
RATIONALE: Giving melphalan and bortezomib before and after a stem cell transplant stops the growth of abnormal cells by stopping them from dividing or killing them. Giving colony-stimulating factors and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy and monoclonal antibody therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This phase II trial is studying how well giving melphalan together with bortezomib followed by stem cell transplant works in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if hematologic responses to high-dose melphalan and autologous stem cell transplantation increase with addition of bortezomib in the conditioning regimen in patients with primary systemic amyloidosis.

OUTLINE:

* Autologous stem cell mobilization and collection: Patients receive filgrastim to mobilize stem cells, which are then collected.
* Conditioning regimen: Patients receive bortezomib intravenously on days -6, -3, 1, and 4 and oral high-dose melphalan on days -2 and -1.
* Stem cell transplantation: Patients undergo autologous stem cell transplantation on day 0.

After completion of study therapy, patients are followed every 6 months for 1 year and annually thereafter.

ELIGIBILITY:
Inclusion criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed primary systemic amyloidosis based on the following criteria:

  * Amyloid light-chain disease
  * Deposition of amyloid material by congo red stain showing characteristic green birefringence
  * Monoclonal light chain protein (Bence Jones protein) in the serum or urine, immunohistochemical studies, or serum free light chain assay
  * Evidence of tissue involvement other than carpal tunnel syndrome (i.e., positive immunohistochemical staining of bone marrow demonstrating clonal plasma cells); tissue amyloid deposits with anti-kappa or anti-lambda anti-serum; evidence for a plasma cell dyscrasia by serum/urine or bone marrow; or overwhelmingly convincing clinical features (e.g., macroglossia) associated with other systemic manifestations

PATIENT CHARACTERISTICS:

* Southwest Oncology Group performance status 0-1
* Fertile patients must use effective contraception
* Left ventricular ejection fraction ≥ 45% by Echocardiogram within the past 60 days
* diffusion capacity of lung for carbon monoxide ≥ 50%

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy with alkylating agent allowed provided there is no morphological or cytogenetic evidence of myelodysplastic syndromes
* Prior total cumulative dose of oral melphalan < 300 mg
* At least 4 weeks since prior cytotoxic therapy and fully recovered

Exclusion criteria:

* No senile, secondary, localized, dialysis-related, or familial amyloidosis
* No overt multiple myeloma (> 30% of bone marrow plasmacytosis, extensive [> 2] lytic lesions, or hypercalcemia)
* Not pregnant or nursing
* No myocardial infarction within the past 6 months, congestive heart failure, or arrhythmia refractory to therapy
* No prior malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer currently in complete remission
  * Any cancer from which the patient has been disease-free ≥ 5 years
* No advanced (grade 3-4) pre-existing neuropathy
* No HIV positivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SCT With Bortezomib and Melphalan: Mobilization with Filgrastim Stem Cell Collection (SCC) Bortezomib Melphalan Stem Cell infusion
  filgrastim: 16 mcg/kg daily beginning 3 days before SCC through day before final SCC
  bortezomib: 1.0 mg/m2/dose D -6, D-3, D +1, D + 4
  melphalan: 100 mg/m2/dose D -2, D -1
  Stem Cell Infusion: infusion of previously collected autologous stem cells
Period: Overall Study
Arm/Group | SCT With Bortezomib and Melphalan
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | SCT With Bortezomib and Melphalan
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematologic Response
Description: complete and partial hematologic response defined as: Complete response: absence of detectable monoclonal protein in serum and urine, and bone marrow biopsy <5% plasma cells with no clonal predominance of kappa or lambda isotype.
  Partial response: any one of the following
  1. For patients with detectable and quantifiable marrow plasmacytosis, a reduction of 50% or more in plasma cells as a percentage of nucleated bone marrow cells.
  2. For patients with a detectable monoclonal peak on serum protein electropheresis or urine protein electropheresis, a reduction in the peak height of 50% or more.
  3. For patients with quantifiable urinary kappa or lambda chain concentration, a reduction in daily light chain excretion (concentration x 24-hr urine volume).
Time Frame: one year
Measure: Number; unit: participants
Groups:
- Stem Cell Transplant With Bortezomib and Melphalan: Mobilization with Filgrastim Stem Cell Collection Bortezomib Melphalan Stem Cell infusion
  filgrastim: 16 mcg/kg daily beginning 3 days before Stem Cell Collectionthrough day before final Stem Cell Collection
  bortezomib: 1.0 mg/m2/dose D -6, D-3, D +1, D + 4
  melphalan: 100 mg/m2/dose D -2, D -1
  Stem Cell Infusion: infusion of previously collected autologous stem cells
Arm/Group | Stem Cell Transplant With Bortezomib and Melphalan
Number analyzed (Participants) | 9
participants | 6

2. Secondary Outcome: Number of Participants Surviving at 100 Days From Transplant
Time Frame: 100 Days from transplant date
Measure: Number; unit: participants
Arm/Group | Stem Cell Transplant With Bortezomib and Melphalan
Number analyzed (Participants) | 9
participants | 9

3. Secondary Outcome: Number of Participants Surviving at 1 Year
Time Frame: one year from transplant
Measure: Number; unit: participants
Groups:
- Stem Cell Transplantation With Bortezomib and Melphalan: Mobilization with Filgrastim Stem Cell Collection Bortezomib Melphalan Stem Cell infusion
  filgrastim: 16 mcg/kg daily beginning 3 days before Stem Cell Collection through day before final Stem Cell Collection
  bortezomib: 1.0 mg/m2/dose D -6, D-3, D +1, D + 4
  melphalan: 100 mg/m2/dose D -2, D -1
  Stem Cell Infusion: infusion of previously collected autologous stem cells
Arm/Group | Stem Cell Transplantation With Bortezomib and Melphalan
Number analyzed (Participants) | 9
participants | 9

4. Secondary Outcome: Number of Participants Surviving at 2 Years
Time Frame: 2 years from transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Transplant With Bortezomib and Melphalan
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | SCT With Bortezomib and Melphalan
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCT With Bortezomib and Melphalan (N=9)
pancytopenia (Blood and lymphatic system disorders) | 9 (9)
coagulation (Blood and lymphatic system disorders) | 1 (1) — fibrinogen
fatigue (General disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
vomit (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3)
heartburn (Gastrointestinal disorders) | 1 (1)
elevated troponin I (Cardiac disorders) | 1 (1)
edema (General disorders) | 2 (2) — limbs
deconditioning (General disorders) | 1 (1)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pneumonia
increased alkylase phosphate (Investigations) | 1 (1)
creatinine increased (Investigations) | 1 (1)
decreased phosphate (Investigations) | 1 (1)
hypocalcemia (Investigations) | 3 (3)
hypoalbuminemia (Investigations) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCT With Bortezomib and Melphalan (N=9)
nausea (Gastrointestinal disorders) | 3 (5)
diarrhea (Gastrointestinal disorders) | 4 (6)
fatigue (General disorders) | 7 (7)
creatinine increased (Investigations) | 1 (1)
deconditioning (General disorders) | 6 (6)
increased alkylase phosphate (Investigations) | 8 (8)
hypocalcemia (Investigations) | 3 (4)
hypoalbuminemia (Investigations) | 1 (1)
hiccups (General disorders) | 4 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes